CLINICAL TRIAL: NCT01579526
Title: A Randomized, Single Dose Study to Determine the Safety and Pharmacokinetics of FP01 Lozenges in Healthy Volunteers
Brief Title: A Single Dose Study to Determine the Safety and Pharmacokinetics of FP01 Lozenges in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Clin01-001
Record Dates: First submitted 2012-04-06; First posted 2012-04-18 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Safety and Pharmacokinetics of FP01 in Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- FP01 Dose 1 (Experimental): Drug
  Interventions: Drug: FP01
- FP01 Dose 2 (Experimental): Drug
  Interventions: Drug: FP01
- FP01 Dose 3 (Experimental): Drug
  Interventions: Drug: FP01
- Comparator (Active Comparator): Drug
  Interventions: Drug: FP01

INTERVENTIONS:
Drug: FP01 — comparison of different dosages

SUMMARY:
The purpose of this study is to determine the safety and pharmacokinetics of FP01 in healthy volunteers.

ELIGIBILITY:
INCLUSION CRITERIA

1. Subjects are male and female volunteers 18 to 55 years of age inclusive.
2. BMI between 18 and 30, inclusive.
3. Subjects must have an estimated creatinine clearance rate of ≥ 80 mL/min as determined by the Cockcroft-Gault equation (see section 7.1).
4. Female subjects of childbearing potential must be using adequate birth control as determined by the Investigator.
5. Female subjects of childbearing potential must have negative pregnancy test results at screening and Day -1.
6. Subjects must be able to provide informed consent after risks and benefits have been explained.
7. Subjects must be non-smoking and non-tobacco user (defined as a subject who has not smoked or used tobacco products for ≥ 12 months from study screening), and must agree to abstain from alcohol and caffeine for 72 hours prior to study dosing and during their participation in the study.
8. Subjects must have a 12 lead ECG without any clinically significant abnormalities of rate, rhythm, intervals or conduction, as determined by the Investigator.
9. Subjects are in generally good health, based on pre-study medical history, physical examination and routine laboratory tests, as determined by the Investigator.
10. Subjects who have no clinically significant disease and/or clinically significant abnormal laboratory values as determined by the Investigator based on medical history, physical examination, or laboratory evaluations conducted at the screening visit or on admission to the clinic.
11. Be willing and able to comply with the study protocol requirements for the duration of the study, including pharmacokinetic sampling

EXCLUSION CRITERIA

1. Females who are pregnant or lactating.
2. Subjects who have a history of drug or alcohol abuse within 12 months of study screening, as determined by the Investigator.
3. Subjects who have participated in any investigational trial within 30 days or six half-lives of the test drug's biologic activity, whichever is longer, before the start of the study (time of first dose).
4. Subjects who have clinically significant medical or psychiatric illnesses currently or within 30 days of start of study (time of first dose), as determined by the Investigator.
5. Subjects with any oral lesions observed at screening visit or at the Day -1 visit.
6. Subjects who have a history of significant allergies (including history of asthma, food, or drug allergies), as determined by the Investigator.
7. Subjects who have had significant blood loss, or have donated or received one or more pints of blood within 30 days prior to dosing.
8. Subjects who have had symptoms of any significant acute illness including upper respiratory infections within 30 days prior to the start of study (time of first dose), as determined by the Investigator.
9. Subjects who have any condition that interferes with their ability to understand or comply with the requirements of the study.
10. Subjects who have a positive drug screen or alcohol screen at study screening or Day -1.
11. Subjects who have any disease or condition (medical or surgical) that might compromise hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or central nervous system function; or any other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the study drug, or that would place the subject at increased risk, as determined by the Investigator.
12. Subjects who have a positive result at screening for HIV, Hepatitis B, or Hepatitis C.
13. Subjects who have received any concomitant prescription, over-the-counter, or herbal medications 7 days prior to study dosing, with the exception of hormonal contraceptives and up to 3 doses of acetaminophen at a dose of 1 gram or less from the time of study screening to the time of study dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic profiles of the active pharmaceutical ingredient | various timepoints over 72 hours
  Plasma PK profiles: various PK indices including, but not limited to, peak plasma concentration (Cmax), Area under the plasma concentration versus time curve (AUC), and elimination half-life (T1/2), and time to peak plasma concentration (Tmax).
Safety and Tolerability | Various Timepoints over 72 Hours
  Safety and Tolerability will take into account the recorded AEs, vital signs, and clinical and laboratory assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Prism Research, Saint Paul, Minnesota, United States